CLINICAL TRIAL: NCT06703801
Title: Evaluation of the Progression of Disease and Health-related Quality of Life in Patients With Pulmonary Hypertension: A Local Clinic-based Registry
Status: Enrolling by invitation | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, GuangMing Tan, assistant professor, Chinese University of Hong Kong
Other Study IDs: 2024.290
Record Dates: First submitted 2024-11-20; First posted 2024-11-25 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Pulmonary Hypertension
Keywords: Pulmonary Hypertension; Six-minute walking test; NT-proBNP
MeSH Terms: conditions — Hypertension, Pulmonary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients at the Prince of Wales Hospital ambulatory cardiac clinic: Patients age > 18 with echocardiographic confirmation of increased pulmonary pressure (eg. estimated RVSP >40mmHg, evidence of RV dilatation etc) and able to attend at the Prince of Wales Hospital ambulatory cardiac clinic

SUMMARY:
Pulmonary Hypertension (PH) is a multifaceted disease and is associated with significant morbidity and mortality if untreated1. Diagnosing PH can be challenging and often delayed2. Multiple international registries included REVEAL3 and COMPERA4 have all demonstrated that diagnostic delay and suboptimal treatment prescription led poor 1 year-survival in patient with PH. In recent years, significant progress has been made in diagnosing, risk stratification, and treatment for patients with PH1. A dedicated PH service has been established in ambulatory clinic to streamline the management of these complex patients. This registry therefore aims to investigate the progression disease and its impact on the quality of life (QoL) of the patients who are managed at the dedicated PH clinic.

DETAILED DESCRIPTION:
Pulmonary Hypertension (PH) is a multifaceted disease and is associated with significant morbidity and mortality if untreated1. Diagnosing PH can be challenging and often delayed2. Multiple international registries included REVEAL3 and COMPERA4 have all demonstrated that diagnostic delay and suboptimal treatment prescription led poor 1 year-survival in patient with PH. In recent years, significant progress has been made in diagnosing, risk stratification, and treatment for patients with PH1. A dedicated PH service has been established in ambulatory clinic to streamline the management of these complex patients. This registry therefore aims to investigate the progression disease and its impact on the quality of life (QoL) of the patients who are managed at the dedicated PH clinic.

ELIGIBILITY:
Inclusion Criteria:

* Patients age > 18 with echocardiographic confirmation of increased pulmonary pressure (eg. estimated RVSP >40mmHg, evidence of RV dilatation etc), and no apparent reversible causes.
* Patients with reasonable pre-morbids and is able to attend ambulatory clinic.

Exclusion Criteria:

* Inability to provide valid consent by the patient or his legal guardian

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with echocardiographic confirmation of increased pulmonary pressure referred for evaluation and management of PH at the Prince of Wales Hospital ambulatory cardiac clinic will be recruited into this registry. Patients' consent will be sought from either the patients or their legal guardian should the patients deemed incapable to consent.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-11-05 (Actual); Primary Completion 2029-11-05 (Estimated); Study Completion 2030-02-05 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality | 3-monthly
  All-cause mortality
WHO functional class | 3-monthly
  Change in functional class (class I as the mildest to class IV as more severe) as measured by WHO functional class over times
EMPASIS-10 questionnaires | 3-monthly
  Change in disease-specific health-related quality of life (QoL) as measured by EMPASIS-10 questionnaires which is an independent prognostic marker in patients with (I/D/H)PAH or CTD-PAH
pulmonary hypertension related mortality | 3-monthly
  pulmonary hypertension related mortality
Borg Rating of perceived exertion (RPE) scale | 3-monthly
  Change in disease-specific health-related quality of life (QoL) as measured by Borg RPE scale which is an outcome measure scale used to gauge one's exercise intensity without the need to rely on physiological parameters
The 5-level EQ-5D version (EQ-5D-5L) | 3-monthly
  Change in disease-specific health-related quality of life (QoL) as measured by EQ-5D-5L which is for assessing patient health states for clinical and economic appraisal
The Modified Medical Research Council (mMRC) Dyspnea scale | 3-monthly
  Change in disease-specific health-related quality of life (QoL) as measured by mMRC which use to access stratifies severity of dyspnea in respiratory diseases, particularly COPD
Pulmonary Embolism Quality of Life Questionnaire (PEmb-QoL) | 3-monthly
  Change in disease-specific health-related quality of life (QoL) as measured by PEmb-QoL which use to access QoL following PE

SECONDARY OUTCOMES:
physical parameters | 3-monthly
  Change in physical parameters
daily activity level | 3-monthly
  Change in daily activity level
Natriuretic Peptide Tests (NT-proBNP) level | 3-monthly
  Change from baseline in log-transformed NT-proBNP level over time
Six-minute walking test (6MWT) | 3-monthly
  Change in Six-minute walking test (6MWT)
Right Ventricular Systolic Pressure (RVSP) as echocardiographic parameters | 3-monthly
  Change in RVSP as echocardiographic parameters
hemodynamic parameters | 3-monthly
  Change in hemodynamic parameters
PH specific medications number and dosage | 3-monthly
  Change of PH specific medications number and dosage over time, including PDE5 inhibitor, Guanyl Cyclase stimulator, Endothelin Receptor antagonist, prostacyclin receptor agonist, and inhaled prostacyclin.
costs of all services, medications and tests | 3-monthly
  The costs of all services, medications and tests as estimated with reference to the Hong Kong Government Gazette 2020 and Hong Kong Hospital Authority Drug Formulary 2020
clinical parameters | 3-monthly
  Change in physical parameters
laboratory parameters | 3-monthly
  Change in laboratory parameters

CONTACTS AND LOCATIONS:
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong, Hong Kong, Hong Kong